CLINICAL TRIAL: NCT01343602
Title: Enhancing Participation of Chronic Stroke Patients in Primary Care by Modified Constraint Induced Movement Therapy (HOMECIMT)
Brief Title: Enhancing Participation of Chronic Stroke Patients by Constraint Induced Movement Therapy (HOMECIMT)
Acronym: HOMECIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMBF-01-GX-1003
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Stroke
Keywords: stroke; Constraint Induced Movement Therapy; participation; Physical Therapy; Occupational Therapy
MeSH Terms: conditions — Stroke | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mod. Constraint-Induced Movement Therapy (Experimental): CIMT at home is applied in the patients' home over the course of four weeks including (i.e. 20 consecutive days) 2 hours of daily training together with an instructed non-professional coach (e.g. family member) applying shaping techniques.
  Interventions: Behavioral: mod. Constraint-Induced Movement Therapy
- Therapy as usual (Other): Patients in this arm will receive usual care dose-matched to the intervention group (250-300 minutes).
  Interventions: Other: Therapy as usual

INTERVENTIONS:
Behavioral: mod. Constraint-Induced Movement Therapy — Therapists of the intervention group are trained in "CIMT at home". During an initial home visit the therapist determines together with the patient an individually tailored home training program focussing on everyday practice and instructs the non-professional coach. For four weeks the patients will perform 2 hours of daily training at home together with an instructed non-professional coach (e.g. family member) applying shaping techniques (i.e. 20 consecutive days). Patients are supposed to wear a resting hand splint for the entire treatment period for 4 to 6 hours daily. During the four weeks the therapist will provide 5 weekly visits at the patients' home to instruct and supervise the training.
  Arms: mod. Constraint-Induced Movement Therapy
Other: Therapy as usual — Therapy as usual consists of the therapy, which is usually provided by the occupational or physical therapist. Therapy will be applied at the patients home or at the therapists' practice.
  Arms: Therapy as usual

SUMMARY:
The aim of this study is to evaluate the efficacy of a modified approach of constraint induced movement therapy ("CIMT at home") for chronic stroke patients, compared to conventional physiotherapy and occupational therapy ("therapy as usual) with regard to the ability to participate in everyday activities.

DETAILED DESCRIPTION:
The study is a parallel cluster randomized controlled trial with therapy practices as clusters. After written consent from the patients, the therapists are randomly assigned to treat either the intervention or the control group. Blinded external assessors evaluate the patients using standardized outcome measures before and after the intervention, and six months later. The two coprimary endpoint assessments of arm and hand function as prerequisites for participation (defined as equal involvement in activities of daily living) are quality of arm and hand use and arm and hand function. Assessments are made four weeks post-treatment and relativized to baseline performance. Changes in primary outcomes are analyzed with mixed models, which consider the hierarchical structure of the data, adjusted to the baseline measurements and sex. The primary analysis compares the two randomized groups, with respect to the adjusted averages for each of the two coprimary endpoints. To keep an overall significance level of 5%, the two endpoints are tested at the significance level of 5% each in hierarchical order.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Stroke onset > 6 months prior to study enrollment
* upper extremity hemiparesis with impairment of hand and/or arm
* minimal function of the hand (at least 10º active wrist extension, at least 10º active of thumb abduction/extension, and at least 10º of extension two additional fingers)
* non-professional coach (e.g. family member)
* prescription of physical or occupational therapy

Exclusion Criteria:

* lack of knowledge of German
* serious impairment of verbal communication ability (e.g. severe aphasia)
* inability to consent (e.g. dementia)
* severe neuro-cognitive deficits (MMSE <23)
* terminal illness, life-threatening co-morbidity
* simultaneous participation in another treatment study targeting stroke recovery
* subjects may not have already received constraint induced movement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Motor Activity Log - Quality Of Movement (MAL-QOM) and Wolf Motor Function Test - Performance Time (WMFT-PT) | 4 weeks (post-treatment) relative to baseline performance
  "Participation" defined as equal involvement in all aspects of society and daily living for people with disabilities is a composite outcome of the following two measures: The MAL-QOM is a self-administered measure of how well 30 daily activities are performed to assess the change in the quality of arm and hand use and the WMFT-PT, measured as the average time (in seconds) to complete 15 tasks, to evaluate the change in arm and hand function.

SECONDARY OUTCOMES:
Motor Activity Log - Quality Of Movement (MAL-QOM) and MAL- Amount Of Use (MAL-AOU) | 3 and 6 months relative to baseline performance
  to assess the change in the quality and amount of arm and hand use
Wolf Motor Function Test - Performance Time (WMFT-PT) and WMFT Functional Ability (WMFT-FA) | 6 months relative to baseline performance
  to assess the change in time and quality of movement
Nine-Hole Peg-Test | 4 weeks (post-treatment) and 6 months relative to baseline performance
  to assess finger dexterity
Stroke-Impact-Scale (SIS) | 4 weeks (post-treatment) and 6 months relative to baseline performance
  to assess the impact on health and quality of life. A self-administered 59-item questionnaire, which assesses 8 domains of stroke (Strength, Hand Function, Activities of Daily Living / Instrumental Activities of Daily Living, Mobility, Communication, Emotion, Memory and Thinking, and Participation)
Barthel Index(BI) | 4 weeks (post-treatment) and 6 months relative to baseline performance
  to assess functional disability i.e. to which somebody can function independently and has mobility in their activities of daily living (ADL)
Instrumental Activities of Daily Living Scale (IADL) | 4 weeks (post-treatment) and 6 months relative to baseline performance
  to asses self-maintaining and instrumental activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Anne Barzel, MD, Principal Investigator — Department of Primary Medical Care, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Primary Medical Care, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Barzel A, Ketels G, Stark A, Tetzlaff B, Daubmann A, Wegscheider K, van den Bussche H, Scherer M. Home-based constraint-induced movement therapy for patients with upper limb dysfunction after stroke (HOMECIMT): a cluster-randomised, controlled trial. Lancet Neurol. 2015 Sep;14(9):893-902. doi: 10.1016/S1474-4422(15)00147-7. Epub 2015 Jul 28. PMID 26231624
- [Derived] Barzel A, Ketels G, Tetzlaff B, Kruger H, Haevernick K, Daubmann A, Wegscheider K, Scherer M. Enhancing activities of daily living of chronic stroke patients in primary health care by modified constraint-induced movement therapy (HOMECIMT): study protocol for a cluster randomized controlled trial. Trials. 2013 Oct 14;14:334. doi: 10.1186/1745-6215-14-334. PMID 24124993